CLINICAL TRIAL: NCT06848972
Title: Development of Exercise Training Programme for Older People with Musculoskeletal Pain in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Islamic University Malaysia (Other)
Responsible Party: Principal Investigator, Nurin Syafiqah binti Mohd Jaias, Principal Investigator, International Islamic University Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIUM/504/14/11/2 IREC2020-KON2
Record Dates: First submitted 2025-02-18; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Musculoskeletal Pain
Keywords: older people; musculoskeletal pain; quality of life; Exercise training programme
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): intervention session, the researcher conducted a structured musculoskeletal exercise programme in the intervention group,
  Interventions: Other: Structured musculoskeletal exercise programme

INTERVENTIONS:
Other: Structured musculoskeletal exercise programme — The module emphasizes specific exercises, strength training with and without weight, flexibility exercises and balancing exercises.

SUMMARY:
The rate of musculoskeletal pain among older people is increasing worldwide and significantly impacts the quality of life. Regular exercise can help prevent and manage chronic musculoskeletal pain because older individuals who are not physically active may have less muscle strength and a higher risk of impairment and injury than physically active persons. As a result, a tailored exercise program may prevent the loss of health-related quality of life among diverse elderly. This study aimed to develop a structured exercise module and identify its effect on musculoskeletal pain and the quality of life of older adults.

DETAILED DESCRIPTION:
Background: The rate of musculoskeletal pain among older people is increasing worldwide and significantly impacts the quality of life. Regular exercise can help prevent and manage chronic musculoskeletal pain because older individuals who are not physically active may have less muscle strength and a higher risk of impairment and injury than physically active persons. As a result, a tailored exercise program may prevent the loss of health-related quality of life among diverse elderly.

Objectives: This study aimed to develop a structured exercise module and identify its effect on musculoskeletal pain and the quality of life of older adults.

Method: A quasi-experimental study was conducted among 60 older adults who experienced musculoskeletal pain in the East Coast Malaysia; Pahang, Terengganu, and Kelantan between January and February 2021. A set of questionnaires contained three parts; Part A: Socio-demographic Background, Part B: Musculoskeletal Pain (Pain Score), and Part C: Functional Limitation. Data was collected using a self-administered questionnaire through an online survey. Data collection processes go through three phases. Phase I: pre-intervention phase, Phase II: intervention session, and Phase III: post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged 60 years old and above
* Lives in East Malaysia; Pahang, Kelantan, and Terengganu
* Have the mental capacity to give informed consent
* Had musculoskeletal pain

Exclusion Criteria:

* Had severely impaired hearing and sight that may have affected their ability to use the self-report scales
* Had neurological diseases or cognitive impairment
* Had a recent self-reported history of stroke or major surgery (in the past 6 months).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Musculoskeletal Pain (Pain Score) | From enrollment to the end of treatment at 6 weeks
  It assess the severity of musculoskeletal pain in older people by using the Numerical Rating Scale (NRS). It ranged from 0 to 10; 0 indicates no pain, 5 for moderate pain, and 10 indicates the worst pain.
Functional Limitation | From enrollment to the end of treatment at 6 weeks
  It focuses on the potential of participants to conduct daily life tasks through the use of the Malay edition of Lawton's Daily Living Instrumental Activities (Kadar et al., 2018; Morrow, 1999). This section includes 8 questions which were based on dichotomous questions (Yes or No). The total possible score is 8. This segment asks about the ability to use the telephone, shop, prepare food, do housekeeping, wash, mode of transport, be responsible of their medication, and their ability in managing their money.

CONTACTS AND LOCATIONS:
Locations (1):
- Pusat Aktiviti Warga Emas (PAWE), Kuantan, Pahang, Malaysia

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available due to confidential issues

REFERENCES:
- [Background] Morrow, S. (1999). Instrumental activities of daily living scale. American Journal of Nursing, 99(1), 24CC.
- [Background] Kadar M, Ibrahim S, Razaob NA, Chai SC, Harun D. Validity and reliability of a Malay version of the Lawton instrumental activities of daily living scale among the Malay speaking elderly in Malaysia. Aust Occup Ther J. 2018 Feb;65(1):63-68. doi: 10.1111/1440-1630.12441. Epub 2018 Jan 9. PMID 29315609